CLINICAL TRIAL: NCT05577936
Title: A Randomized Controlled Trial of the Next Science® XPERIENCE™ Advanced Surgical Irrigation Versus Standard of Care Irrigation Efficacy in Decreasing Bioburden in Primary Total Hip and Knee Arthroplasty Wounds
Brief Title: Xperience™ vs Normal Saline Irrigation Solution for Decreasing Bioburden After Primary Total Hip and Knee Arthroplasty
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Delay in funding.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Cameron K. Ledford, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-004244
Record Dates: First submitted 2022-10-09; First posted 2022-10-13 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Total Knee Replacement Surgery; Total Hip Replacement Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Xperience no rinse antimicrobial solution group (Experimental): XPERIENCE Advanced Surgical Irrigation will be utilized as the final wash after the TKA or THA procedure prior to closure
  Interventions: Device: XPERIENCE Advanced Surgical Irrigation
- Normal saline solution group (Active Comparator): Standard of care irrigation will be utilized as the final wash after the TKA or THA procedure prior to closure.
  Interventions: Other: Standard of Care Irrigation

INTERVENTIONS:
Device: XPERIENCE Advanced Surgical Irrigation — A clear, colorless, aqueous solution that is indicated for use in the cleansing and removal of debris, including microorganisms, from wounds. Soak for 3 minutes for a total volume of 1L
  Arms: Xperience no rinse antimicrobial solution group
Other: Standard of Care Irrigation — 17.5 mL povidone-iodine with 500 mL normal saline: solution (0.35%) for 3 minutes for a total volume of 1L (including a normal saline rinse)
  Arms: Normal saline solution group

SUMMARY:
The purpose of this study is to evaluate the effectiveness of Xperience, a no rinse antimicrobial solution, on joint infection rates in patients undergoing total hip (THA) and total knee (TKA) arthoplasty surgery.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo primary total hip (via direct anterior approach, press-fit components) or total knee arthroplasty (via manual approach, cemented components).
* Willing to comply with all study-related procedures and be available for the duration of the study.
* Provide signed and dated informed consent.

Exclusion Criteria:

* Unable to provide signed and dated informed consent.
* Unwilling or unable to comply with all study-related procedures.
* Known history of sensitivity or allergic reaction to any of the study products or its components, including any products used for standard of care (such as dressings or any coverings).
* Has underlying condition or state that, in the 'investigator's opinion, would make them too critically ill to complete the day 90 postoperative follow ups.
* Pregnant, planning to become pregnant, or nursing female subjects.
* Subject with any mental impairment or condition that would make them unable to properly consent without use of LAR or additional subject protections.
* Subject is a prisoner and/or part of a vulnerable subject population, which necessitates additional human research subject protections beyond the scope of this protocol.
* Subject with an active infection or systemic antibiotic therapy within 2 weeks prior to surgery with the exception of preoperative antimicrobial prophylaxis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in culture positive rates | Baseline (pre-irrigation) and post-irrigation approximately 3 minutes
  Number of culture positive tissue samples

SECONDARY OUTCOMES:
Deep Periprosthetic Joint Infection | 90 days
  Number of subjects to have deep periprosthetic joint infection within 90 days of index operation

CONTACTS AND LOCATIONS:
Overall Officials: Cameron Ledford, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials